CLINICAL TRIAL: NCT02906215
Title: Mobile Application to Improve Care Coordination Among HIV Clinic and Substance Use Treatment Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Kasey Claborn, Assistant Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R34DA041237 (NIH)
Record Dates: First submitted 2016-08-23; First posted 2016-09-20 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: HIV; Substance Use; Care Coordination
Keywords: mHealth; implementation; PrEP; digital health
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Care Coordination Intervention (Experimental): The care coordination intervention will consist of a mobile application designed for treatment providers, an interagency communication protocol, and a series of cross-training in HIV and addiction issues.
  Interventions: Behavioral: Care Coordination Intervention

INTERVENTIONS:
Behavioral: Care Coordination Intervention — cross-training in HIV/PrEP and substance use, plus a digital health tool to improve evidence-based screening, brief intervention, referral to treatment, and patient management across HIV, PrEP, and addiction treatment providers

SUMMARY:
Many people living with HIV use illicit drugs and require treatment for both HIV and drug use, however, many barriers exist which prevent integration of dual care services. This study will develop a novel intervention aimed at the provider-level which will combine an evidence-based training model with use of mobile technology to improve care coordination between providers at HIV clinics and substance use treatment facilities. If proven effective, this intervention may be widely disseminated and easily implemented into existing clinic structures, thereby improving care coordination among providers and linkage to dual treatment for HIV-infected people who use drugs.

DETAILED DESCRIPTION:
Drug use is associated with poor linkages to HIV care, reduced retention in care, increased sexual risk behavior, and decreased adherence to medications, leading to inferior clinical outcomes, and increased HIV transmission. HIV-infected people who use drugs (HPWUD) have higher rates of co-occurring psychiatric and medical diagnoses, resulting in increased utilization of services. Many structural and systemic barriers impede the integration of treatment for HIV and substance use (SU). The use of a mobile application combined with an evidence-based training model offers an innovative approach to improving care coordination and linking patients to care in need of dual treatment. A mhealth application delivered via tablet device provides a unique channel to link HIV and SU treatment providers located at off-site clinics. This study will be a Stage I pilot and feasibility study that will be the first to use a theory-based model of care coordination to develop a Care Coordination Intervention (CCI) for treatment providers serving HPWUD. This study seeks to develop a secure mobile technology platform that will: (a) enable rapid communication among providers at multiple clinics, (b) improve linkage to dual care, and (c) improve coordination of patient services. The CCI will also utilize an evidence-based training model to increase provider knowledge in relevant HIV, PrEP, and SU issues. The proposed method of integrating dual care for patients is expected to be an efficient and easily disseminable platform for integrating HIV/SU care that will facilitate communication between providers at multiple clinics and allow for efficient management of patient treatment referrals and service utilization. This project will examine acceptability, feasibility, and sustainability potential using mixed-methods. A three-phase, top-down research approach to adapt, refine, and pilot test the intervention will be conducted. Phase 1 will include individual interviews with key stakeholders and audits of referral and communication processes within each clinic. Phase 2 will include development of the CCI. The investigators will conduct a functionality test and conduct a series of interviews with key stakeholders to inform iterative revision of the CCI. During Phase 3, the investigators will train providers in the CCI and evaluate the feasibility, acceptability, and sustainability potential among HIV and SU treatment providers located at two different clinics via a pre-, post-test design. Data will be gathered at the organizational-, provider-, and patient-levels. Compared to pre-implementation of the CCI in both clinics, the investigators expect that post-implementation data will result in: (H1) greater satisfaction of care coordination at the provider level; (H2) increased frequency and improved quality of interagency communications; (H3) enhanced interagency professional relationships; and (H4) increased dual care retention at the patient level. The long-term goal is to expand the availability of sustainable interventions to improve coordination of HIV and SU treatment services. Data from this research will form the basis of a future multisite R01 proposal for this early career, new investigator applicant.

ELIGIBILITY:
Inclusion Criteria:

* Participants must:

  * be at least 18 years of age,
  * provide either HIV care or substance abuse treatment [e.g., physicians, residents, psychologists, mid-level providers],
  * be employed at a participating recruitment site, and (d) able to provide informed consent.

Exclusion Criteria:

* Physical impairments that prevent completion of the intervention, cognitive impairments that jeopardize informed consent, active psychosis, and not fluent in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Interagency Collaboration as measured by the "Levels of Collaboration" scale | 1-, 3-, and 6-months

SECONDARY OUTCOMES:
Acceptability of the Care Coordination Intervention | 6-months
  Acceptability will assessed using satisfaction ratings.
Usability of the Mobile Application | 6-months
  Usability will be assessed through quantifying online usage patterns.
Change in frequency and quantity of communication | 1-, 3-, and 6-months
  Data will be extracted through the online dashboard to examine change in communication between providers at the two participating clinics.
Provider Perception Inventory will assess change in provider-related stigma | 1-, 3-, and 6-months
  This questionnaire measures health service providers' stigma in regards to HIV, substance use, and sexual risk behavior.
Implementation Climate Scale | Baseline
  This scale will measure the degree to which there is a strategic organizational climate supportive of the intervention implementation in each participating clinic.
Change in Patient Treatment Retention in both HIV and Substance Use Services | 1-, 3-, and 6-months
  Data will be extracted through the online dashboard to examine change in appointment attendance for patients enrolled in treatment at the participating HIV and substance use clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Kasey Claborn, PhD, Principal Investigator — The University of Texas
Locations (1):
- The University of Texas Dell Medical School, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Claborn K, Becker S, Ramsey S, Rich J, Friedmann PD. Mobile technology intervention to improve care coordination between HIV and substance use treatment providers: development, training, and evaluation protocol. Addict Sci Clin Pract. 2017 Mar 14;12(1):8. doi: 10.1186/s13722-017-0073-1. PMID 28288678